CLINICAL TRIAL: NCT07233226
Title: Role of Hyaluronic Acid in Type I Tympanoplasty for Total and Subtotal Tympanic Membrane Perforations
Brief Title: Role of Hyaluronic Acid Gel as an Adjunct to Temporalis Facia Graft in Tympanoplasty for Total Tympanic Membrane Perforation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hemdan, Assistant Professor of Otorhinolaryngology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.22.01.1835
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Tympanoplasty
Keywords: hyaluronic acid gel; tympanoplasty; total tympanic membrane perforation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia (Experimental)
  Interventions: Procedure: Tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia
- Tympanoplasty using temporalis fascia (Experimental)
  Interventions: Procedure: Tympanoplasty using temporalis fascia

INTERVENTIONS:
Procedure: Tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia — Underlay tympanoplasty through postauricular approach using hyaluronic acid gel that will be added to the temporalis fascia graft as well as the perforation edges
  Arms: Tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia
Procedure: Tympanoplasty using temporalis fascia — Underlay tympanoplasty through postauricular approach using temporalis fascia
  Arms: Tympanoplasty using temporalis fascia

SUMMARY:
Aim: the aim of the study is to compare the results of tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia graft with tympanoplasty using temporalis fascia graft.

Study Design: A prospective single blinded randomized controlled trial that will be carried out on 60 cases with total tympanic membrane perforation who will undergo tympanoplasty at our tertiary referral center. All involved cases will have grade IV tympanic membrane perforation based on Saliba classification for tympanic membrane perforation.

The patients will be randomly divided into 2 groups A and B. Patients in group A will undergo underlay tympanoplasty using temporalis fascia graft with the utilization of hyaluronic acid gel was used as an adjunct to temporalis fascia graft. Patients in group B will undergo classic underlay tympanoplasty using temporalis fascia graft.

The two group will be compared as regards:

1. Graft success rate.
2. Hearing outcome
3. Surgical complications

DETAILED DESCRIPTION:
Aim: the aim of the study is to compare the results of tympanoplasty using hyaluronic acid gel as an adjunct to temporalis fascia graft with tympanoplasty using temporalis fascia graft.

Study Design: A prospective single blinded randomized controlled trial that will be carried out on 60 cases with total tympanic membrane perforation who will undergo tympanoplasty at our tertiary referral center. Prior to study conduction, institutional ethics committee approval was obtained (code: MS.19.04.576). Informed written consents well be obtained from all cases before surgeries.

All involved cases will have grade IV tympanic membrane perforation based on Saliba classification for tympanic membrane perforation where the perforation was total perforation involving the entire four quadrants of the tympanic membrane. All the cases will have inactive dry ear for at least 2 months prior to surgeries. All involved cases will be ≥18 years old. Excluded cases include revision cases, cases with active (discharging ear), cases < 18 years old, immunocompromised cases and cases who missed to follow up.

The patients will be randomly divided into 2 groups A and B using computer generated block randomization. Patients in group A will undergo underlay tympanoplasty using temporalis fascia graft through postauricular approach with the utilization of hyaluronic acid gel was used as an adjunct to temporalis fascia graft. Patients in group B will undergo classic underlay tympanoplasty using temporalis fascia graft through postauricular approach.

The two group will be compared as regards:

1. Graft success rate.
2. Hearing outcome
3. Surgical complications

ELIGIBILITY:
Inclusion Criteria:

* Grade IV tympanic membrane perforation based on Saliba classification for tympanic membrane perforation.
* Inactive dry ear for at least 2 months prior to surgeries.

Exclusion Criteria:

* Revision cases.
* Cases who missed to follow up.
* Cases with active (discharging) ear.
* Immunocompromised cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Graft success | 6 months
  Prescence of an intact non-retracted tympanic membrane

SECONDARY OUTCOMES:
Hearing improvement | 6 months
  Reduction of postoperative mean air conduction threshold and air bone gap in comparison to the preoperative results

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology Department, Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt